CLINICAL TRIAL: NCT05899868
Title: Utilization of Airway Stabilizing Rod to Assist With LMA Guided Fiberoptic Intubation in Children
Brief Title: Utilization of Airway Stabilizing Rod
Acronym: FASTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Arvind Chandrakantan, Associate Professor of Anesthesiology, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: H50120
Record Dates: First submitted 2023-05-16; First posted 2023-06-12 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Airway Complication of Anesthesia

STUDY DESIGN:
Intervention Model Description: Testing of device for success during endotracheal intubation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Time to intubation using FASTER device (Other): Time from fiberoptic placement into airway to documentation of end-tidal carbon dioxide waveform through the endotracheal tube.
  Interventions: Device: Time to Intubation using FASTER device

INTERVENTIONS:
Device: Time to Intubation using FASTER device — Time from fiberoptic placement onto airway to documentation of end-tidal carbon dioxide waveform through the endotracheal tube.
  Other Names: FASTER

SUMMARY:
The pediatric airway is known to be more challenging than the adult airway when performing endotracheal intubation. When a patient cannot be ventilated and/or intubated, the guidelines for airway management dictate that a laryngeal mask airway (LMA) be used as a rescue device to oxygenate and ventilate the patient. While an excellent device the LMA is seen as temporary and ultimately needs to be replaced by an endotracheal tube (ETT).

DETAILED DESCRIPTION:
The objective is to study this device in patients with difficult airway to assess the success rate and time to intubation for placing an endotracheal tube using this device.

ELIGIBILITY:
Inclusion Criteria:

* Ages 5-18 years
* Requiring intubation
* Known difficult airway
* LMA placement possible

Exclusion Criteria:

* Known normal airway
* Procedure not requiring endotracheal intubation
* Parental refusal
* Patient dissent

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Overall time in the airway | 5 minutes
  Time from fiberoptic placement onto airway to documentation of end-tidal carbon dioxide waveform through the endotracheal tube.
Total time to intubation | 3 minutes
  Time from movement of the device to documentation of end-tidal carbon dioxide waveform through the endotracheal tube.

CONTACTS AND LOCATIONS:
Overall Officials: Arvind Chandrakantan, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hosppital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
This pilot data will not be shared

REFERENCES:
- [Derived] Adler AC, Duong K, Chandrakantan A. Fiberoptic-Assisted Endotracheal Rod for Endotracheal Intubation Through a Supraglottic Airway in Patients with Difficult Intubation: A Clinical Device Study. Anesth Analg. 2025 Apr 1;140(4):986-989. doi: 10.1213/ANE.0000000000007268. Epub 2024 Nov 21. No abstract available. PMID 39774053